CLINICAL TRIAL: NCT04455451
Title: Intensive Care Therapy of Covid-19 Disease in Germany an Multi-center Observational Study
Brief Title: Intensive Care Therapy of Covid-19 Disease in Germany
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: DCIR
Record Dates: First submitted 2020-07-01; First posted 2020-07-02 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-09

CONDITIONS: COVID; ARDS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multi-center retrospective and prospective observational study of Covid-19 patients with severe or critical illness treated on a German ICU

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* Covid-19 disease (positive SARS-CoV-2 PCR)

Exclusion Criteria:

-none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults admitted for ICU therapy due to severe or critical Covid-19
Sampling Method: Non-Probability Sample
Enrollment: 2054 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Mortality | up to 150 days
  ICU Mortality of patients

SECONDARY OUTCOMES:
ICU length of stay | up to 150 days
  Intensive care unit length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rosenberger, MD, PhD, Principal Investigator — University Hospital Tübingen; Harry Magunia, MD, Principal Investigator — University Hospital Tübingen
Locations (27):
- Germany (27):
  - RWTH Aachen - Department for operative Intensive Care Medicine and intermediate Care, Aachen
  - Zollernalbklinikum, Balingen
  - Charité Universitätsmedizin Berlin, Berlin
  - UH Bochum - Department for Anesthesiology and Intensive Care Medicine, Bochum
  - Universitätsklinikum Bonn, Bonn
  - Klinikum der Universität Witten/Herdecke - Köln / Klinik für Anästhesiologie und operative Intensivmedizin, Cologne
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Ev. Krankenhaus Bethesda Duisburg Klinik für Anästhesiologie und Intensivmedizin, Duisburg
  - Univerrsitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Frankfurt, Frankfurt
  - University Hospital Freiburg - Department for Anesthesiology and Intensive Care Medicine, Freiburg im Breisgau
  - Universitätsklinikum Giessen Klinik für Anaesthesiologie und operative Intensivmedizin, Giessen
  - Universitätsmedizin Göttingen Klinik für Anästhesiologie, Göttingen
  - Universitätsklinikum Greifswald, Greifswald
  - Universitätsklinikum Halle, Halle
  - University Hospital Heidelberg - Department for Anesthesiologie and Intensive Care Medicine, Heidelberg
  - Universitätsklinikum des Saarlandes, Homburg/Saar
  - Universitätsklinikum Leipzig, Leipzig
  - UKSH Campus Lübeck - Department for Anesthesiology and Intensive Care Medicine, Lübeck
  - University Hospital Magdeburg - Department for Anesthesiology and Intensive Care Medicine, Magdeburg
  - Universitätsklinikum Marburg, Marburg
  - Technische Universität München, München
  - Oberschwabenklinik Ravensburg Klinik für Anästhesie-, Intensiv-, Notfall- und Schmerzmedizin, Ravensburg
  - University Hospital Tübingen - Department for Anesthesiology and Intensive Care Medicine, Tübingen
  - Universitätsklinikum Ulm, Ulm
  - Universitätsklinikum Würzburg Klinik und Poliklinik für Anästhesiologie, Intensivmedizin und Schmerztherapie, Würzburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Magunia H, Lederer S, Verbuecheln R, Gilot BJ, Koeppen M, Haeberle HA, Mirakaj V, Hofmann P, Marx G, Bickenbach J, Nohe B, Lay M, Spies C, Edel A, Schiefenhovel F, Rahmel T, Putensen C, Sellmann T, Koch T, Brandenburger T, Kindgen-Milles D, Brenner T, Berger M, Zacharowski K, Adam E, Posch M, Moerer O, Scheer CS, Sedding D, Weigand MA, Fichtner F, Nau C, Pratsch F, Wiesmann T, Koch C, Schneider G, Lahmer T, Straub A, Meiser A, Weiss M, Jungwirth B, Wappler F, Meybohm P, Herrmann J, Malek N, Kohlbacher O, Biergans S, Rosenberger P. Machine learning identifies ICU outcome predictors in a multicenter COVID-19 cohort. Crit Care. 2021 Aug 17;25(1):295. doi: 10.1186/s13054-021-03720-4. PMID 34404458
- See also: Study Landing Page — https://www.medizin.uni-tuebingen.de/de/covid-intensivstudie